CLINICAL TRIAL: NCT04660266
Title: Accuracy of Ultrasound Exam, Including Doppler and Elastography, in the Diagnosis of VOD, in the 21 Days Following Bone Marrow Transplantation
Brief Title: Accuracy of Ultrasound Exam, Including Doppler and Elastography, in the Diagnosis of VOD, Following Bone Marrow Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0696-20-RMB
Record Dates: First submitted 2020-11-18; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: VOD; Ultrasound Therapy; Complications

STUDY DESIGN:
Intervention Model Description: liver evaluation by US before, 14 days and 21 days after bone marrow transplantation, in the purpose to predict the appearance of Veno occlusive disease.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all cohort (Other)
  Interventions: Diagnostic Test: Liver Ultrasound

INTERVENTIONS:
Diagnostic Test: Liver Ultrasound — liver ultrasound examination, including gray-scale and seven Doppler examination

SUMMARY:
The purpose of the study:

Validation of the use of intentional ultrasound examination, which includes Doppler and elastography for the diagnosis of obstructive venous disease of the liver within 21 days after bone marrow transplantation.

Protocol:

Patients who are planned for a bone marrow transplantaion will be recruited for the study by the staff of the Transplant Department. Inclusion criteria: Patients over the age of 18 before a bone marrow transplantation.

Eligibility criteria: Transplanted under 18 years of age

Research protocol:

After informed consent, patients will undergo an ultrasound examination before the transplant.

After 14 days and again after 21 days patients will undergo two more US exams, If there is a change in their clinical condition the patients will undergo additional examination accordingly.

At the same time on the 14th and 21st day a clinical evaluation will be performed by the clinical physician in the transplant department based on clinical criteria of European Blood and Brain Transplant Association (EBMT).

The results of the clinical evaluation and blood test results will be collected.

Patients will be divided into two groups:

* Control group: Patients who did not develop VOD( veno occlusive disease ) during 21 days.
* Study group: Patients who developed VOD during 21 days.

All ultrasound examination data will be compared between the two groups in

In addition will be collected:

* Demographics - age, sex.
* Background diseases including heart and liver diseases.
* Basic disease as a transplantation cause.

All data will be collected anonymously and coded separately.

DETAILED DESCRIPTION:
The purpose of the study:

Validation of the use of intentional ultrasound examination, which includes Doppler and elastography for the diagnosis of obstructive venous disease of the liver within 21 days after bone marrow transplantation.

Protocol:

Patients who are planned for a bone marrow transplantaion will be recruited for the study by the staff of the Transplant Department. Inclusion criteria: Patients over the age of 18 before a bone marrow transplantation.

Eligibility criteria: Transplanted under 18 years of age

Research protocol:

After informed consent, patients will undergo an ultrasound examination before the transplant.

The test will include:

1. Demonstration of liver including its size.
2. Gallbladder demonstration including its width and wall thickness.
3. Main portal vein width, Speed and flow direction in main portal vein.
4. Evaluation of umbilical vein in the falciform ligament to check existence of flow and venous width in case it opened.
5. Assessment of existence a small / medium or large amount of ascites measurement of resistance index in the main hepatic artery.
6. Complete elastography examination.

After 14 days and again after 21 days patients will undergo two more US exams, If there is a change in their clinical condition the patients will undergo additional examination accordingly.

At the same time on the 14th and 21st day a clinical evaluation will be performed by the clinical physician in the transplant department based on clinical criteria of European Blood and Brain Transplant Association (EBMT).

The results of the clinical evaluation and blood test results will be collected.

Patients will be divided into two groups:

* Control group: Patients who did not develop VOD( veno occlusive disease ) during 21 days.
* Study group: Patients who developed VOD during 21 days.

All ultrasound examination data will be compared between the two groups in

In addition will be collected:

* Demographics - age, sex.
* Background diseases including heart and liver diseases.
* Basic disease as a transplantation cause.

All data will be collected anonymously and coded separately.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 before a bone marrow transplantation.

Exclusion Criteria:

* Transplanted under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy of liver ultrasound in predicting VOD | 21 days
  ultrasound results inculding gray scale , doppler and elastography will be compared to the clinical diagnosis of VOD the diagnosis of VOD will be performed according to the Europian Society for Blood and Marrow transplantation revised criteria
  1. presence of ascites yes/no
  2. liver enlagement more than 17 cm
  3. Bilirubin >2 mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israek, Israel

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/6363247/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19766729/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17768390/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/8420443/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/3321587/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27183098/
- See also: Related Info — https://europepmc.org/article/med/30895833
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9240551/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29767845/
- See also: Related Info — https://www.x-mol.com/paper/1276245089442099200